CLINICAL TRIAL: NCT06237673
Title: A Randomized, Controlled Trial in Patients With Suspected Coronary Artery Disease Based on Acute or Chronic Atypical Angina Pectoris - EXTEND
Brief Title: The "CAD-Man" EXTEND Study
Acronym: CAD-Man-EXTEND
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marc Dewey, Prof. Dr. Dr. h.c. Marc Dewey, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EA1/124/23
Record Dates: First submitted 2023-12-20; First posted 2024-02-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT (Experimental): CT-directed clinical management strategy
  Interventions: Diagnostic Test: CT
- Invasive coronary angiography (ICA) (Active Comparator): Standard clinical management directed by conventional invasive coronary angiography (ICA).
  Interventions: Diagnostic Test: invasive coronary angiography (ICA)

INTERVENTIONS:
Diagnostic Test: CT — CT-directed clinical management strategy
  Arms: CT
Diagnostic Test: invasive coronary angiography (ICA) — Standard clinical management directed by conventional invasive coronary angiography (ICA).
  Arms: Invasive coronary angiography (ICA)

SUMMARY:
CAD-Man Extend is the long-term follow-up (clinical, laboratory, and computed tomography (CT) imaging) of a single-center, randomized, controlled CAD-Man trial comparing a CT-first strategy with a direct- invasive coronary angiography (ICA) diagnostic and management strategy, in 329 patients clinically referred for ICA with atypical angina or chest pain.

Overall goal:

The extension of CAD-Man follow-up (clinical, laboratory, and CT imaging) to approximately 10 years will provide the opportunity to compare plaque burden with CT-guided management versus direct-ICA at long-term and other endpoints.

DETAILED DESCRIPTION:
The CAD-Man (Coronary Artery Disease Management with Multislice Computed Tomography and Magnetic Resonance Imaging in Patients with Atypical Angina Pectoris) trial evaluated whether computed tomography (CT) or invasive coronary angiography (ICA) should be performed in patients clinically referred for coronary angiography with an intermediate probability of coronary artery disease. Patients with suspected CAD were randomized 1:1 ratio to CT, followed by ICA if positive for obstructive CAD, or to direct ICA. In both tests, obstructive CAD was defined as at least a 50% diameter stenosis in the left main coronary artery or at least a 70% diameter stenosis in other coronary arteries. Investigators and participants were blinded to randomization sequence but could not be blinded to the assigned group because of the apparent differences between CT and ICA. Independent investigators, who were blinded to the randomization group and were not part of the study team, anonymously assessed outcomes. Results on the comparative effectiveness of CT and ICA in preventing the primary outcome of major procedural complications within 48 hours of the last procedure and major adverse events (defined as cardiovascular death, nonfatal myocardial infarction, or nonfatal stroke) were published for a median follow-up of 3.3 years.

The primary results and additional subgroup analyses of the CAD-Man trial led to three new hypotheses that will be evaluated in the CAD-Man Extend study.

1. Main hypothesis:

   Whether CT-guided management of patients with atypical angina results in a reduction in coronary plaque burden (as determined by repeat CT scan) compared with direct-ICA management until 10 years.
2. Secondary hypothesis:

1. Whether clinical characteristics or blood levels and lipid-lowering medications have an impact on intraindividual progression of coronary plaques in patients in the CT group.

2. Whether primary CT examination in patients with atypical angina leads to a reduction in chronic impairment of renal function after 10-years compared with initial ICA examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected CAD
* Patients with atypical angina
* Patients who have previously participated in the CAD-Man study and have not died at a median follow-up of 3.3 years.

Exclusion Criteria:

Exclusion criteria for additional CT scan:

* Pregnancy
* Any health condition that would cause concern that participation would not be in the best interest of health (eg, extensive comorbidities)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of coronary plaque burden (non-calcified plaque volume (NCPV) measured by CT at 10-years between the initial randomization CT and ICA groups | at 10 years
Comparison of coronary plaque burden total plaque volume (TPV)) measured by CT at 10-years between CT and ICA groups | at 10 years

SECONDARY OUTCOMES:
Intraindividual progression of coronary artery disease (defined as change in coronary plaque burden from the first CT until the CT examination after 10 years) in the CT group. | at 10 years
Comparison of the difference in chronic kidney injury, (eGFR and as increase in creatinine by 25% or 0.5 mg/dl) in both groups at 10-year follow-up between CT and ICA groups. | at 10 years

OTHER OUTCOMES:
To compare minor cardiovascular events at final follow-up (after approximately 10 years). | at 10 years
  Cardiovascular events (unstable angina pectoris, re-revascularization, and first revascularization at least 2 months after randomization)
To compare the cost-effectiveness in both groups. (after 10 years). | at 10 years
  To compare cost-effectiveness in both groups using the quality-adjusted life year data, and cost data derived from the trial.
Comparison of two types of structured reports one medical and one using easy language (according to the german clinical practice guidelines) using patient acceptance questionnaire. | at 10 years
To compare cholesterol level (LDL, HDL, Triglycerin) between the initial randomization CT and ICA groups. | at 10 years
Comparison of statin use (proportion) between the initial randomization CT and ICA groups. | at 10 years
Effect of statins on coronary plaque burden (non-calcified plaque volume (NCPV) )measured by CT at 10-years in CT group | at 10 years
Effect of statins on coronary plaque burden (total plaque volume (TPV)) measured by CT at 10-years in CT group | at 10 years
To compare calcified plaque volume at 10-years between CT and ICA group | at 10 years
To compare low-attenuation plaque volume (LAPV) at 10-years between CT and ICA group | at 10 years
To compare percentage atheroma volume (PAV) at 10-years between CT and ICA group | at 10 years
To compare relative plaque volume at 10-years between CT and ICA group | at 10 years
To compare segment stenosis score (SSS) at 10-years between CT and ICA group | at 10 years
To compare segment involvement score (SIS) at 10-years between CT and ICA group | at 10 years
To compare stenosis at 10-years between CT and ICA group | at 10 years
  Stenosis (no stenosis, <20%, 20 to 50%, >50%)
To compare plaque composition at 10-years between CT and ICA group | at 10 years
  (calcified, non-calcified (fibrous, fibrofatty, lipid-rich), partially calcified)
To compare high-risk plaque (HRP) features at 10-years between CT and ICA group | at 10 years
  (HRP; positive remodelling (PR), napkin ring sign, spotty calcification, low attenuation (LAP)
To analyze the impact of baseline cardiovascular risk factors on non-calcified plaque volume (NCPV) in the CT Group | at 10 years
  Age (< 65, 65-75, > 75)
  Body Mass Index (BMI) (< 25, 25-30, > 30) Gender (male versus female) Diabetes (yes/no)
To analyze the impact of baseline cardiovascular risk factors on total plaque volume (TPV) in the CT Group | at 10 years
  Age (< 65, 65-75, > 75)
  Body Mass Index (BMI) (< 25, 25-30, > 30) Gender (male versus female) Diabetes (yes/no)
To analyze the impact of nutrition on non-calcified plaque volume (NCPV) in the CT Group | at 10 years
To analyze the impact of nutrition on total plaque volume (TPV) in the CT Group | at 10 years
To analyze the impact of physical activity (Freiburg questionnaire) on non-calcified plaque volume (NCPV) in the CT Group | at 10 years
To analyze the impact of physical activity (Freiburg questionnaire) on total plaque volume (TPV) in the CT Group | at 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will share individual patient data from CAD-Man extend study via the GUIDE-IT platform.
Supporting Information: Study Protocol
Time Frame: 12 months after publication. End 3 years after publication
Access Criteria: Researchers who provide a methodologically sound proposal approved by the Dissemination Committee of CAD-Man and GUIDE-IT.
  The study proposal must include: The proposed study's overview, rationale, aims and analysis methods, plans for dissemination of results and names of those wishing to access data, and how is the data going to be stored and for how long.
URL: http://www.guide-it.org

REFERENCES:
- [Background] Dewey M, Rief M, Martus P, Kendziora B, Feger S, Dreger H, Priem S, Knebel F, Bohm M, Schlattmann P, Hamm B, Schonenberger E, Laule M, Zimmermann E. Evaluation of computed tomography in patients with atypical angina or chest pain clinically referred for invasive coronary angiography: randomised controlled trial. BMJ. 2016 Oct 24;355:i5441. doi: 10.1136/bmj.i5441. PMID 27777234
- [Background] Schonenberger E, Martus P, Bosserdt M, Zimmermann E, Tauber R, Laule M, Dewey M. Kidney Injury after Intravenous versus Intra-arterial Contrast Agent in Patients Suspected of Having Coronary Artery Disease: A Randomized Trial. Radiology. 2019 Sep;292(3):664-672. doi: 10.1148/radiol.2019182220. Epub 2019 Jul 2. PMID 31264950
- [Background] Bosserdt M, Martus P, Tauber R, Dreger H, Dewey M, Schonenberger E; CAD-Man Study Group Investigators. Serum creatinine baseline fluctuation and acute kidney injury after intravenous or intra-arterial contrast agent administration-an intraindividual comparison as part of a randomized controlled trial. Nephrol Dial Transplant. 2022 May 25;37(6):1191-1194. doi: 10.1093/ndt/gfac013. No abstract available. PMID 35090035
- [Background] Bosserdt M, Feger S, Rief M, Preuss D, Ibes P, Martus P, Kofoed KF, Laule M, Perez I, Dewey M. Performing Computed Tomography Instead of Invasive Coronary Angiography: Sex Effects in Patients With Suspected CAD. JACC Cardiovasc Imaging. 2020 Mar;13(3):888-889. doi: 10.1016/j.jcmg.2019.10.014. Epub 2019 Dec 18. No abstract available. PMID 31864987
- [Background] Laskowski D, Feger S, Bosserdt M, Zimmermann E, Mohamed M, Kendziora B, Rief M, Dreger H, Estrella M, Dewey M. Detection of relevant extracardiac findings on coronary computed tomography angiography vs. invasive coronary angiography. Eur Radiol. 2022 Jan;32(1):122-131. doi: 10.1007/s00330-021-07967-x. Epub 2021 Jun 15. PMID 34129067
- [Background] Feger S, Elzenbeck L, Rieckmann N, Marek A, Dreger H, Beling M, Zimmermann E, Rief M, Chow BJW, Maurovich-Horvath P, Laule M, Tauber R, Dewey M. Effect of Computed Tomography Versus Invasive Coronary Angiography on Statin Adherence: A Randomized Controlled Trial. JACC Cardiovasc Imaging. 2021 Jul;14(7):1480-1483. doi: 10.1016/j.jcmg.2021.01.032. Epub 2021 May 19. No abstract available. PMID 34023253